CLINICAL TRIAL: NCT06923982
Title: The Effect of Using Virtual Reality Glasses on Post-Care Pain and Comfort Level in Intensive Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çankırı Karatekin University (Other)
Responsible Party: Principal Investigator, Emre Şahin, Specialist Nurse, Çankırı Karatekin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CankırıKU-HEM-ES-01
Record Dates: First submitted 2024-03-21; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Copd; Heart Failure; Intensive Care Unit Syndrome; Renal Failure; Gastro Esophageal Reflux
Keywords: nursing; virtual reality; pain; comfort; intensive care unit
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Renal Insufficiency; Gastroesophageal Reflux; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Two groups were taken as experimental and control groups
Masking Description: In the experimentally planned study, patients diagnosed with cancer hospitalized in the 10-bed internal medicine intensive care unit at Eskişehir Osmangazi University Hospital were first evaluated in terms of the inclusion criteria, and individuals who did not meet the criteria were excluded from the study. Eligible individuals were included in one of the intervention group and control groups using virtual reality glasses by randomization method. The lottery method was used to randomize individuals to research groups. In this method, 30 pieces of red and blue paper were placed into 2 black fabric bags by the researcher. Red paper represents the intervention group and blue paper represents the control group. Individuals who met the inclusion criteria and agreed to participate in the study were asked to randomly choose a piece of paper from the bags. In this way, the groups were automatically balanced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual reality (Other): During care, patients are given a duration of 3-10 minutes. virtual reality glasses (VR box 2.0 virtual glasses) for a total of 15 minutes walks in parks, nature and seaside with music background, with reality glasses (6.5 inches), videos that the patient wants to watch and whenever he/she wants, such as underwater or museum tours. Videos that could be changed were shown.
  Interventions: Other: virtual reality, experimental group; Other: control group

INTERVENTIONS:
Other: virtual reality, experimental group — Socio-demographic characteristics form questions were asked to individuals in the intervention group before care. During the care, patients are given virtual reality glasses (VR box 2.0 virtual reality glasses and 6.5 inch) for a total of 15 minutes, ranging from 3 to 10 minutes, and watch videos that the patient wants to watch, such as park, nature and seaside walks, undersea and museum trips, with a music background. and he was shown videos that he could change at any time. After the maintenance, Visual Analog Scale-Pain (VAS-P) scale, General Comfort Level Scale and Satisfaction Evaluation Scale for Virtual Reality Glasses Application questions were applied. 24 hours after the care, VAS-P and General Comfort Level Scale were administered again.
Other: control group — A socio-demographic questionnaire was administered to the control group before care. During maintenance, no intervention was applied and standard care in routine practice was applied. After the care, Visual Analog Scale-Pain (VAS-P) scale and General Comfort Scale were applied. 24 hours after the treatment, the Visual Analog Scale-Pain (VAS-P) scale and the General Comfort Scale were applied again.

SUMMARY:
The aim of this study is to determine the level of pain and comfort associated with the implementation of virtual reality prior to nursing care in patients undergoing treatment in the intensive care unit. The research will be conducted in the Internal Medicine Intensive Care Unit of a university hospital.

DETAILED DESCRIPTION:
The aim of this study is to determine the level of pain and comfort associated with the implementation of virtual reality prior to nursing care in patients undergoing treatment in the intensive care unit.

The study will be conducted in the Internal Medicine Intensive Care Unit of a university hospital. The study population will consist of patients admitted to the internal medicine unit who are between 18 and 65 years of age, are conscious with a Glasgow Coma Scale (GCS) score of 10 or above, have no auditory or visual impairments, and are not receiving mechanical ventilation support.

A total of 60 patients will be included in the study and randomly assigned into two groups: 30 in the experimental group and 30 in the control group.

Data will be collected through face-to-face interviews using a Sociodemographic Characteristics and Information Description Form, a Visual Analog Scale (VAS), and the General Comfort Scale - Short Form (GCS-SF).

The intervention for the experimental group will include viewing calming videos using a virtual reality headset before nursing care. Pain and general comfort levels will be evaluated 24 hours after the nursing care procedure.

Statistical analyses such as percentage calculations, t-test, Mann-Whitney U test, and Spearman correlation analysis will be used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are hospitalized in the intensive care unit (with diagnoses such as cancer, chronic renal failure, heart failure, gastrointestinal bleeding, COPD, DM, etc.) and volunteer to participate in the study.
* Between the ages of 18-65,
* Having clear consciousness, orientation to place, time and person, and having a GCS score of 10 and above,
* Individuals who do not have any hearing or visual impairment,
* They were determined as individuals who were not on mechanical ventilation support.

Exclusion Criteria:

* Receiving mechanical ventilation support
* Individuals under 18 years of age and over 65 years of age

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in Pain Level Measured by Visual Analog Scale (VAS) Before and After Nursing Care | 24 hours
  Pain will be assessed using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain). Higher scores indicate worse pain. Pain levels will be measured before care and again 24 hours after nursing care, and compared between the experimental and control groups.
Change in Overcoming Problems Sub-dimension and General Comfort Level (GCS-SF) After Virtual Reality Application | 24 hours
  Comfort will be assessed using the General Comfort Scale - Short Form (GCS-SF), including the "overcoming problems" sub-dimension. The GCS-SF total score ranges from 24 to 96, with higher scores indicating greater comfort. Scores will be measured 24 hours after the virtual reality application in both the experimental and control groups.
Change in Refreshment/Comfort Sub-Dimension Scale Score After Virtual Reality Application | 24 hours
  Comfort will be evaluated using the Refreshment/Comfort sub-dimension of the General Comfort Scale - Short Form (GCS-SF). Scores range from 8 to 32, with higher scores indicating greater comfort. Scores will be measured 24 hours after the virtual reality application in both the experimental and control groups.

OTHER OUTCOMES:
Satisfaction Survey Score Related to the Use of Virtual Reality Glasses in the Experimental Group | 24 hours
  Participants in the experimental group will wear virtual reality glasses during nursing care. Their satisfaction will be evaluated through a self-report questionnaire using a scale ranging from 0 (not satisfied at all) to 10 (extremely satisfied). Higher scores indicate greater satisfaction. The survey will be administered 24 hours after the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Çankırı Karatekin Üniversitesi, Çankırı, Turkey (Türkiye)